CLINICAL TRIAL: NCT01114399
Title: Diet and Vascular Health Study
Acronym: BROCCOLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other); University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2009IFR01
Record Dates: First submitted 2010-04-27; First posted 2010-05-03 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Disease; Cardiovascular Disease risk (mild to moderate); Cholesterol; Ambulatory blood pressure; Arterial Stiffness
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Broccoli (Experimental): Standard Broccoli
  Interventions: Dietary Supplement: Diet and Vascular Health
- High Glucosinolate Broccoli (Experimental): High Glucosinolate Broccoli
  Interventions: Dietary Supplement: Diet and Vascular Health
- Peas (Experimental): Peas
  Interventions: Dietary Supplement: Diet and Vascular Health Study

INTERVENTIONS:
Dietary Supplement: Diet and Vascular Health — One group will consume 400g of standard broccoli each week for 12weeks; the second group will consume 400g of the high glucosinolate broccoli each week for 12weeks while the third group will consume 400g of peas each week for 12weeks. The broccoli and the peas will be consumed on top of the volunteer's standard diet.
  Arms: Standard Broccoli
Dietary Supplement: Diet and Vascular Health — One group will consume 400g of standard broccoli each week for 12weeks; the second group will consume 400g of the high glucosinolate broccoli each week for 12weeks while the third group will consume 400g of peas each week for 12weeks. The broccoli and the peas will be consumed on top of the volunteer's standard diet.
  Arms: High Glucosinolate Broccoli
Dietary Supplement: Diet and Vascular Health Study — One group will consume 400g of standard broccoli each week for 12weeks; the second group will consume 400g of the high glucosinolate broccoli each week for 12weeks while the third group will consume 400g of peas each week for 12weeks. The broccoli and the peas will be consumed on top of the volunteer's standard diet.
  Arms: Peas

SUMMARY:
The aim of this study is to examine the effects of a diet rich in broccoli on cardiovascular disease risk using biochemical indicators such as blood lipid profiles, most notably cholesterol; markers of inflammation as well as established physiological measurements such as Pulse wave velocity (PWV), Augmentation index (AIx) and Ambulatory Blood Pressure Measurements (ABPM). Broccoli contains compounds known as glucosinolates which are metabolised to isothiocyanates when consumed. The major glucosinolate in broccoli is known as glucoraphanin which produces the isothiocyanate sulforaphane. The glucosinolates are thought to be the principal component in broccoli that may reduce CVD risk. The investigators will use a standard cultivar of broccoli and a cultivar that has enhanced levels of glucosinolates ('HG broccoli'). This broccoli has been used in previous intervention studies (e.g. ClinicalTrials.gov NCT00535977). Volunteers will be asked to consume 400g of standard broccoli, HG broccoli or peas each week over a 12 week period in a double blinded (for the broccoli) parallel study. The volunteers recruited will, according to the Joint British Societies (JBS 2) Guidelines on the prevention of cardiovascular disease (CVD) in clinical practise, have a 10-20% (mild to moderate) risk of developing cardiovascular disease or having a cardiovascular (CV) event in the next 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 50 years will be recruited onto the study using the JBS 2 cardiac risk assessor calculator (Copyright University of Manchester 1998): Scores of 10-20% will be acceptable for participation in the study.
* Total cholesterol ≥ 5.0mmol/L
* Blood pressure measurements

  * Systolic≥ 120mmHg
  * Diastolic ≥ 80mmHg
  * BMI ≥20
  * Smokers and Non Smokers

Exclusion Criteria:

* Diagnosed diabetics;
* Fasting glucose >6mmol/L;
* Blood pressure <90/50 or 95/55 if symptomatic; >160/100
* Chronic kidney disease;
* Those on any lipid lowering therapies like statins, bile acid sequestrants, cholesterol absorption inhibitors and nicotinic acid;
* Those who have suffered a cardiovascular event like stroke, myocardial infarction or trans ischemic attacks;
* Peripheral vascular disease including Claudication
* Consumption of fish oil supplements (unless volunteer is willing to discontinue their use 4 weeks prior to the start of the)
* Parallel participation in another research project which involves dietary intervention and/or sampling of biological fluids/materials
* Any person related or living with any member of the study team
* Participation in another research project which involves blood sampling within the last four months; Blood from both studies should not exceed 470mL
* BMI <20
* BMI >40
* Fasting total cholesterol > 8.0mmol/L
* Gastrointestinal disease (excluding hiatus hernia) unless symptomatic or study intervention/procedure is contraindicated
* Going on holiday for more than 7 days in any single period or within 2 weeks of their clinical appointment at the CRTU
* Currently suffering from or have suffered from any neck and throat injuries and surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Examination of the indicators of CVD after the consumption of broccoli, high glucosinolate broccoli and peas. | Week 12
  To examine the effects of a diet rich in broccoli on the systemic indicators of CVD including total cholesterol as well as established physiological measurements such as ambulatory blood pressure (BP), Augmentation Index (AIx) and Pulse Wave velocity (PWV) in subjects with a mild to moderate (10-20%) risk of developing CVD within the next 10 years

SECONDARY OUTCOMES:
The determination of key polymorphic genes of the trial subjects | Baseline
  To determine the genotype of individuals for key polymorphic genes (GSTM1, GSTT1 and GSTP1) and relate them to observed changes in CVD risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Armah CN, Traka MH, Dainty JR, Defernez M, Janssens A, Leung W, Doleman JF, Potter JF, Mithen RF. A diet rich in high-glucoraphanin broccoli interacts with genotype to reduce discordance in plasma metabolite profiles by modulating mitochondrial function. Am J Clin Nutr. 2013 Sep;98(3):712-22. doi: 10.3945/ajcn.113.065235. PMID 23964055